CLINICAL TRIAL: NCT05863468
Title: Quantification of the Airflow Into Sinuses Before and After ArchSinus Implantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: STS Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 461010P
Record Dates: First submitted 2023-01-29; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-01

CONDITIONS: Chronic Sinusitis, Ethmoidal

STUDY DESIGN:
Intervention Model Description: 4 chronic sinusitis patients will undergo unilateral or bilateral in-office middle turbinate medialization and subsequent ArchSinus implantation. Baseline and 12-week airflow rate and particle deposition will be analyzed with Computational Modeling Analysis. symptomatic improvement will be analyzed using SNOT-22 and NOSE questioners.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ArchSinus implantation (Experimental): Subjects will undergo unilateral or bilateral in-office middle turbinate medialization and subsequent ArchSinus implantation
  Interventions: Device: ArchSinus implantation

INTERVENTIONS:
Device: ArchSinus implantation — Unilateral or bilateral in-office middle turbinate medialization and subsequent ArchSinus implantation

SUMMARY:
This is a single-center, single-arm, interventional case study designed to compare the sinonasal airflow and symptomatic status of four (4) chronic sinusitis patients, before and after the ArchSinus stent implantation.

DETAILED DESCRIPTION:
This is a single-center, single-arm, interventional case study. This case study is designed to compare the sinonasal airflow and symptomatic status of four (4) chronic sinusitis patients who after undergoing primary FESS were seen to have symptomatic lateralization of the middle turbinate and underwent medialization of the middle turbinate accompanied by ArchSinus stent implantation.

Patient eligibility will be confirmed based on the endoscopic examination and SNOT-22 score.

Patient history will be taken, specifically which if any nasal spacer was used after the primary FESS.

4 chronic sinusitis patients that suffer from middle turbinate lateralization and symptomatic deterioration, 3-6 months after primary FESS, that met the inclusion / exclusion criteria, will undergo unilateral or bilateral in-office middle turbinate medialization and subsequent ArchSinus implantation. The stents will be removed 2-3 weeks after procedure.

CT scan will be performed at baseline and 12 weeks after the ArchSinus stent removal, and 3D sinonasal airways reconstruction of the maxillary, ethmoid, sphenoid & frontal sinuses will be performed. Subsequently, airflow and particle deposition will be simulated in each reconstruction, and airflow rate and particle deposition will be quantified for different sinuses.

Symptomatic status will be analyzed at baseline and 1, 6 and 12 weeks after the ArchSinus stent removal using SNOT-22 and NOSE Questioners.

Debridement is disallowed during the ArchSinus implantation time period. Nasal decongestions are disallowed prior to CT scan examination.

ELIGIBILITY:
Inclusion Criteria:

* Male/female, 18 year or older
* Diagnosis of chronic rhinosinusitis defined as symptomatic inflammation of the sinuses of at least 12 consecutive weeks duration despite medical management
* ≥ 3 months post primary FESS
* Symptoms of chronic rhinosinusitis defined as ≥ 10 score on SNOT-22
* Middle turbinate lateralization defined as ˃ 2 score on MT lateralization scale

Exclusion Criteria:

* Polyp grade ˃ 4 bilaterally on Lildholdt's scale (1-3)
* Sinonasal tumors
* Known allergy to nickel
* Known polyurethane induced dermatitis
* History of immune deficiency
* Cystic fibrosis
* Pregnant or lactating female
* Acute sinus inflammation
* Coagulation disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Estimated)
Dates: Start 2023-06-15 (Estimated); Primary Completion 2023-11-21 (Estimated); Study Completion 2023-12-21 (Estimated)

PRIMARY OUTCOMES:
Sinus airflow and particle deposition rate | 12 weeks
  The primary objective of this study aims to compare the sinonasal airflow rate and particle deposition rate at Baseline and 12 weeks after the ArchSinus stent implantation, based on CFD analysis.

SECONDARY OUTCOMES:
Symptomatic improvement | 12 weeks
  The secondary objective of this study is to analyze correlation between an increased sinus airflow and symptomatic improvement, assessed using SNOT-22 and NOSE Questioners, at baseline and at 1, 6 and 12 weeks after the ArchSinus stent removal.

IPD SHARING:
Plan to Share IPD: No